CLINICAL TRIAL: NCT05051410
Title: Effect of Intracanal Cryotherapy on Postoperative Pain Using Two Different Irrigation Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Maryam Rafique, principal investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRafique
Record Dates: First submitted 2021-09-03; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
Keywords: cryotherapy; postoperative pain; single visit; negative pressure irrigation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: subject are randomly placed into one of the three groups:control,intracanal cryotherapy with needle irrigation, intracanal cryotherapy with EndoVac system. cold saline will be used in intracanal cryotherapy for five minutes. postoperative pain will be evaluated for 7 days using visual analogue scale.
Who Masked: Participant, Outcomes Assessor
Masking Description: it is doubled blinded study in which participants will be blinded. the assessor, who will assess the postoperative pain of participant will also be blinded regarding the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control (No Intervention): single visit root canal treatment will be performed with no additional irrigation.
- intracanal cryotherapy with needle irrigation (Experimental): single visit root canal treatment will be performed with additional irrigation with cold saline using needle irrigation.
  Interventions: Procedure: intracanal cryotherapy using needle irrigation and EndoVac system
- intracanal cryotherapy using Endovac system (Experimental): single visit root canal treatment will be performed with additional irrigation with cold saline using EndoVac system.
  Interventions: Procedure: intracanal cryotherapy using needle irrigation and EndoVac system

INTERVENTIONS:
Procedure: intracanal cryotherapy using needle irrigation and EndoVac system — a cold saline will be used as final irrigant in two groups but with different irrigation systems.
  Arms: intracanal cryotherapy using Endovac system; intracanal cryotherapy with needle irrigation

SUMMARY:
this study was conducted to know the effect of intracanal cryotherapy on postoperative pain using two different irrigation systems to deliver the cold saline.

method: A total of 75 patients presenting with a diagnosis of irreversible pulpitis with symptomatic apical periodontitis in single rooted teeth were included in the study and randomly divided into three groups (n=25) (i.e. Control group, cryotherapy group with needle irrigation and cryotherapy group with negative pressure irrigation system). After complete root canal cleaning and shaping, final irrigation was done with 2.5°c 0.9% physiological saline in cryotherapy groups with needle irrigation (NI) and negative pressure irrigation system (NPI) whereas in control group no additional irrigation was done. Root canal treatment was completed in single visit. Participants were asked through telephone to rate their postoperative pain intensity after root canal treatment by visual analogue scale from day 1 till day 7 on given proforma.

two way repeated measures of ANOVA test were applied to know the mean difference between and among the groups.

DETAILED DESCRIPTION:
Intracanal cryotherapy is one of the methods recently used to reduce the postoperative pain. The aim of this randomized control trial was to evaluate the effect of cold saline (cryotherapy) as a final irrigant on postoperative pain with two different irrigation systems after single visit root canal treatment objective: To find out the effect of cryotherapy as a final irrigant after root canal preparation on postoperative pain using needle irrigation and negative pressure irrigation system (EndoVac).

method: the intervention used in this study was intracanal cryotherapy with two different irrigation systems i.e. needle irrigation and negative pressure irrigation system(EndoVac). for cryotherapy cold saline was used at temperature of 2.5 °c. total sample size was calculated was 75 by using PASS version 11.non probability purposive sampling was used for patient recruitment. three groups were made with sample size of 25 in each group. group allocation was done by computer generated random numbers.according to inclusion and exclusion criteria patients were selected and after complete diagnosis patients were thoroughly explained about the treatment and informed consent were taken. to record the preoperative pain ,patients were provided a proforma. proforma consisted of visual analogue scale for pain record. endodontic procedure was performed by the principal investigator and it was same in all the three groups.final irrigation protocol was diferent among the groups; control group:no final irrigation was done, cryotherapy with needle irrigation: with needle irrigation cold saline was delivered,cryotherapy with EndoVac: with EndoVac cold saline was delivered. obturation in root canal was done with same protocol in all the groups.and access cavity was filled with temporary restoration. postoperative instruction was given to the patient and follow up procedure has also been explained to them. follow up was consisted of 7 days and through phone call by assessor which was blind regarding the groups. at day 7, patient were returned with proforma in which they have noted the pain score of 7 days and at the same visit temporary filling was replaced by permanent one. the principal investigator was blind regarding the postoperative pain,as it was done by some other assessor.

statistical analysis was done by using SPSS v.16.the two-way ANOVA repeated measures was performed for mean comparision among and between the groups.chi-square/fischer exact test test was performed for analgesic intake.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years.
* No significant present and past medical findings.
* Mature, single rooted teeth with single canal and closed apices.
* Symptomatic irreversible pulpitis with symptomatic apical periodontitis (moderate to severe pain according to VAS).
* Periodontal status- healthy periodontium according to Classification of Periodontal Disease and Conditions. (i.e. code 0).

Exclusion Criteria:

* Immature teeth with open apices.
* Root presenting with resorption, fracture, root caries, root curvature ≥ 10°.
* Calcified canals.
* Pregnancy.
* systemic disorders and taking medications
* Perio - endo lesion

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
incidence of postoperavtive pain after intracanal crytherapy using two different irrigation systems | post operative pain was assessed for 7 days after treatment,visual analogue scale was used to assess the pain
  visual analogue scale (VAS) was used to assess postoperative pain after the treatment.Proforma was provided to the patient which include VAS. The scale is usually a 10 cm line with clearly defined boundaries. 0= no pain,1-3=mild pain,4-6=moderate pain and 7-10=severe pain.patient marked the number according to their pain level..

CONTACTS AND LOCATIONS:
Overall Officials: Maryam rafique, MDS, Principal Investigator — DUHS
Locations (1):
- Maryam rafique, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No